CLINICAL TRIAL: NCT02169700
Title: Ischemic Compression After Dry Needling of a Latent Myofascial Trigger Point Reduces Post-needling Soreness Intensity and Duration.
Brief Title: Ischemic Compression on Post-needling Soreness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, PhD, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10/2014
Record Dates: First submitted 2014-06-17; First posted 2014-06-23 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Neck Pain
Keywords: Ischemic compression; Myofascial trigger points; Post-needling soreness
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ischemic compression. Dry Needling (Experimental): Ischemic compression was carried out after dry needling.
  Interventions: Procedure: Ischemic compression. Dry Needling
- Sham Ischemic compression. Dry Needling (Sham Comparator): Sham Ischemic compression was carried out after dry needling.
  Interventions: Procedure: Ischemic compression. Dry Needling
- Control group (No Intervention): No intervention. Control group

INTERVENTIONS:
Procedure: Ischemic compression. Dry Needling — Ischemic compression was carried out after dry needling. Dry needling was performed with a solid filament needle. Subjects were asked to lie in a prone position. The MTrP was held firmly in a pincer grasp. Before inserting the needle, the patient was advised about the possible sharp pain and muscle twitching. The needle was inserted perpendicular to the skin. Then, the muscle fibers were repeatedly perforated by rapidly inserting and partially withdrawing the needles from the MTrP until two local twitch responses were elicited from the muscle. On removal of the needle, the area was compressed firmly with a cotton bud for two minutes. Immediately after the needling, subjects were randomly assigned to one of three groups (IC, sham and control).
  Arms: Ischemic compression. Dry Needling; Sham Ischemic compression. Dry Needling

SUMMARY:
Myofascial trigger points (MTrPs) are identified through physical examination as hypersensitive spots within taut bands of skeletal muscle, painful on compression, triggering characteristic referred pain and generating motor dysfunction as well as autonomic phenomena. Different dry needling procedures have been described in the treatment of MTrPs. Needling therapies which consist in partially inserting and withdrawing the needle from the trigger point site in order to elicit local twitch responses are associated with higher effectiveness in releasing MTrPs. Deep dry needling has obtained a grade A recommendation compared to sham, for immediate reduction of pain in patients with upper-quadrant myofascial pain syndrome. Nevertheless, trigger point dry needling are frequently associated to a post-needling soreness. The application of ischemic compression (IC) after trigger point injection in the upper trapezius muscle has shown higher reduction of pain and disability in myofascial pain patients, compared with trigger point injection alone. To the authors' knowledge, no previous studies have evaluated the effectiveness of IC or any manual therapy methods for the treatment of post-needling soreness. The aims of this study were: (a) to evaluate the effectiveness of IC on reducing post-needling soreness after dry needling of one latent MTrP in the upper trapezius muscle, and (b) to investigate the effect dry needling combined with IC, compared to dry needling alone and dry needling combined with placebo IC will have on cervical range of motion (c) to determine whether psychological factors are predictive of postneedling pain and (d) to analyze if the relationships between psychological variables and postneedling pain varied as a function of postneedling soreness treatment

ELIGIBILITY:
Inclusion Criteria:

* Subjects were included if they presented at least one latent MTrP in the upper trapezius muscle

Exclusion Criteria:

* Presence of coagulation disorders
* Neck or facial pain
* Previous application of a dry needling technique
* MTrP therapy in head or neck within the previous 3 months
* Fibromyalgia
* An insurmountable fear of needles as a reason of refusing the treatment
* History of surgery in the head or neck area

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2013-12; Primary Completion 2014-02 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | From Baseline in pain intensity at during needling and at 72 hours
  VAS. Despite being a subjective evaluation, it has been documented in previous studies its reliability and validity and its sensitivity to the clinical changes. For this reason, this scale has been used in numerous clinical trials. The patient places a vertical mark on a flat horizontal line of 10 cm. One extreme is 0 (no pain) and the other extreme is 10 (maximum pain) and it must be a difference of 2 points in the evaluation range to produce minimal improvement which is clinically significant

SECONDARY OUTCOMES:
Cervical Range of Motion (CROM) | CROM measurements were taken before needling, after the intervention, and at 24 and 72 hours post-treatment.
  The subjects sat in a chair and a CROM goniometerc was placed over his or her head. They were asked to perform active neck movements to the fullest extent of their mobility. Each movement was recorded three times and the average value was calculated. The CROM measurement device has proven to be a reliable measure33 of movement, with an intra-rater reliability ranging from 0.7 to 0.9 and an inter-rater reliability ranging from 0.8 to 0.87.

OTHER OUTCOMES:
Psychological variables | Before dry needling intervention
  Catastrophizing, kinesiophobia, pain anxiety and fear of pain

CONTACTS AND LOCATIONS:
Overall Officials: Josué Fernández Carnero, PhD, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

REFERENCES:
- [Derived] Martin-Pintado-Zugasti A, Pecos-Martin D, Rodriguez-Fernandez AL, Alguacil-Diego IM, Portillo-Aceituno A, Gallego-Izquierdo T, Fernandez-Carnero J. Ischemic Compression After Dry Needling of a Latent Myofascial Trigger Point Reduces Postneedling Soreness Intensity and Duration. PM R. 2015 Oct;7(10):1026-1034. doi: 10.1016/j.pmrj.2015.03.021. Epub 2015 Mar 31. PMID 25836591